CLINICAL TRIAL: NCT02167113
Title: Collection of Plasma Samples From Individuals Initiating Therapy With Entecavir or Tenofovir for Chronic Hepatitis B Virus Infection for the Clinical Evaluation of the Aptima HBV Quant Assay
Brief Title: Collection of Samples for the Clinical Evaluation of the Aptima HBV (Hepatitis B Virus) Quant (Quantification) Assay
Acronym: HBVQuant
Status: Completed | Type: Observational
Sponsor: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: V10434-HBVQPS-CSP-01; V10434-HBVQPS-CSP-01 (Other: Hologic)
Record Dates: First submitted 2014-06-12; First posted 2014-06-18 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study population

SUMMARY:
This non-interventional clinical study will be conducted to prospectively collect serial plasma samples from subjects with chronic HBV infection who are initiating antiviral therapy. These samples will be used to estimate clinical utility endpoints for the Aptima HBV Quant assay, which is used as an aid in the management of HBV-infected patients undergoing HBV antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject is chronically infected with HBV.The subject is treatment naïve and is initiating HBV antiviral therapy with either entecavir or tenofovir as indicated in the FDA approved label
* The subject will be considered treatment naïve if he/she had <12 weeks of oral antiviral therapy with any nucleoside or nucleotide therapy
* The subject is at least 18 years of age at the time of enrollment
* Adequate medical records are available for collection of protocol-defined demographics, baseline patient characteristics, medical history, virology and specific laboratory results, and other information to verify enrollment criteria
* The subject and/or legally authorized representative is willing and able to provide consent prior to providing a specimen(s)

Exclusion Criteria:

* Subject is in one of the following patient populations:

  * Acute HBV infection
  * Patients who are HBV immune tolerant
  * Human immunodeficiency virus (HIV) and/or hepatitis C virus (HCV) co-infection
  * Solid organ or bone marrow transplant recipients
  * Renal failure or dialysis
  * Evidence or history of hepatic decompensation
  * Evidence or history of hepatocellular carcinoma
* Underlying liver disease other than HBV
* Receiving chemotherapy, immunosuppressive agents
* Subject is unsuitable for study participation based on the Investigator's decision (eg, unlikely to comply with study visit schedule, significant medical complication)
* Participating in another investigational study that the Investigator believes might interfere with the subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment naïve men and women ≥18 years of age with chronic HBV infection initiating entecavir or tenofovir treatment.
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
Association between virologic response at Week 12 (assessed using the Aptima HBV Quant assay) and virologic response at Week 48 (assessed using an FDA-approved HBV quant assay). | Week 48 (from start of therapy)
  Virologic response is defined as HBV DNA levels less than the lower limit of quantitation at the assessed time point.
  Association will be measured as an odds ratio.
Association between virologic response at Week 24 (assessed using the Aptima HBV Quant assay) and virologic response at Week 48 (assessed using an FDA-approved HBV quant assay). | Week 48 (from start of therapy)
  Virologic response is defined as HBV DNA levels less than the lower limit of quantitation at the assessed time point.
  Association will be measured as an odds ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Kuslich, Study Director — Hologic, Inc.
Locations (88):
- United States (38):
  - Banner Health Good Samaritan, Phoenix, Arizona
  - Dignity Health - St. Joseph's Hospital, Phoenix, Arizona
  - Advanced Rx Clinical Research, Garden Grove, California
  - High Desert Gastroenterology, Lancaster, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Inland Empire Liver Foundation, Rialto, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Foundation Hospital, San Francisco, California
  - San Jose Gastroenterology, San Jose, California
  - South Bay Gastroenterology Medical Group, Torrance, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Schiff Center for Liver Disease, Miami, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - The Research Institute, Springfield, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Sing Chan, MD, Flushing, New York
  - North Shore University Hospital, Manhasset, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Piedmont HealthCare, Statesville, North Carolina
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Austin Center for Clinical Research, Austin, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Harborview Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Australia (3):
  - Napean Hospital, Gastroenterology and Hepatology Department, Kingswood, New South Wales
  - Liverpool Hospital, Department of Gastroenterology, Sydney, New South Wales
  - St Vincent's Hospital Department of Gastroenterology, Fitzroy, Victoria
- Bulgaria (3):
  - UMHAT Dr. Gerogi Stranski, Clinic of Gastroenterology, Pleven
  - UMHAT Aleksandrovska, Clinic of Gastroenterology, Sofia
  - UMHAT Sveti Ivan Rilski Clinic of Gastroenterology, Sofia
- Canada (6):
  - Foothills Medical Centre, Calgary, Alberta
  - Lair Centre, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Toronto Liver Centre, Toronto, Ontario
- Germany (8):
  - Leberzentrum am Checkpoint Fachärztegemeinschaft für innere Krankheiten, Berlin
  - Medizinische Klinik mit Schwerpunkt Hepatologie und Gastroenterologie, Berlin
  - Zentrum für Infektiologie Berlin Prenzlauer Berg, Berlin
  - Universitätsklinikum Essen Klinik für Gastroenterologie und Hepatologie, Essen
  - ifi-Studien und Projekte GmbH An der Asklepios Klinik St. Georg, Haus L, Hamburg
  - ifi-Studien und Projekte GmbH, An der Asklepios Klinik St. Georg, Hamburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsmedizin Mannheim II. Medizinische Klinik, Mannheim
- Hungary (4):
  - Szent István és Szent László Kórház, Budapest
  - Budai Hepatollógiai Központ, Budapest
  - Szent János Kórház, Budapest
  - Pándy Kálmán Megyei Kórház, Gyula
- Italy (3):
  - 'Ospdale Da Procida, Salerno
  - 'Medicina Interna - Ospedale Civile, Sassari
  - Medicina Interna - Ospedale Civile, Sassari
- New Zealand (3):
  - Auckland Liver Research Unit, Grafton, Auckland
  - Waikato Gastroenterology and Respiratory Research Office, Hamilton West, Waikato Region
  - Gastroenterology Research, Wellington Hospital, Newton, Wellington Region
- Romania (7):
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Sector 1, București
  - Institutul de Boli Infectioase "Prof. Dr. Matei Bals", Sector 2, București
  - Institutul Clinic Fundeni, Bucuresti, Sector 2, București
  - Spitalul Universitar de Urgenta Bucuresti, Sector 5, București
  - Spitalul Clininc de Boli Infecţioase Constanţa, Constanța, Constanța County
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu, Jud. Sibiu
  - Policlinica Algomed, Timisoara, Timișoara, Jud. Timis
- Turkey (Türkiye) (13):
  - Istanbul University Cerrahpaşa School of Medicine, Istanbul, Istanbul
  - Ankara University School of Medicine, Ankara
  - Yıldırım Beyazıt University Atatürk Training and Research Hospital, Ankara
  - Adnan Menderes Üniversitesi, Aydin
  - Uludag University School of Medicine, Bursa
  - Dicle University School of Medicine, Diyarbakır
  - Osmangazi University School of Medicine, Eskişehir
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Dokuz Eylül University School of Medicine, Izmir
  - Kocaeli University School of Medicine, Kocaeli
  - Selçuk University School of Medicine, Konya
  - Ondokuz Mayıs University School of Medicine, Samsun
  - Karadeniz Technical University School of Medicine, Trabzon